CLINICAL TRIAL: NCT00576238
Title: A Multi Centre, Parallel, Randomised Study of the Skin Tolerance of Betamethasone Creams on Atopic Eczema and the Influence of Moisturiser Treatment on the Recurrence of Eczema
Brief Title: Skin Tolerance Study of Betamethasone Creams in Atopic Eczema and the Preventative Properties of a Moisturiser
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACO Hud Nordic AB (Industry)
Responsible Party: Berit Berne, Hudkliniken, Akademiska sjukhuset, Uppsala
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ACO/02/08
Record Dates: First submitted 2007-12-18; First posted 2007-12-19 (Estimated); Last update posted 2008-10-13 (Estimated); Status verified 2008-10

CONDITIONS: Atopic Eczema
Keywords: Atopic eczema; Topical corticosteroid
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Betamethasone Valerate; Urea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1:1 (Experimental): Part 1 - eczema treatment
  Interventions: Drug: betamethasone valerate
- 1:2 (Active Comparator): Part 1 - eczema treatment
  Interventions: Drug: betamethasone valerate
- 2:1 (Experimental): Part 2 - maintenance treatment
  Interventions: Drug: urea
- 2:2 (No Intervention): Part 2 - maintenance treatment

INTERVENTIONS:
Drug: betamethasone valerate — Topical application according to a fixed schedule for three weeks
  Other Names: Betnoderm 0,1 % kräm
  Arms: 1:1
Drug: betamethasone valerate — Topical application according to a fixed schedule for three weeks
  Other Names: Betnovat kräm 0,1%
  Arms: 1:2
Drug: urea — Topical application twice daily for up to 6 months
  Other Names: Canoderm kräm 5%
  Arms: 2:1

SUMMARY:
Topical steroid creams as well as moisturizing creams are important parts of the treatment strategy of atopic eczema. This study aims to investigate the tolerance of a new strong steroid cream in comparison to an already marketed reference cream with equal amount of active but with different cream vehicle. The second part of the study will investigate the possible preventative property of a moisturizing cream on skin that has been previously cleared from eczema.

ELIGIBILITY:
Inclusion Criteria:

* Females and males between 18 and 65 years of age
* Caucasian
* AD according to the criteria of Hanifin and Rajka (12) with eczematous lesions corresponding to an Atopic Dermatitis Severity Index (ADSI) (13) score of at least 6 on any of the following areas: arms, legs, chest, abdomen or back
* No serious health conditions that may interfere with the study
* Written informed consent

Exclusion Criteria:

* Eczematous regions exclusively in intertriginous areas or in the face
* Use of topical steroids or any other dermatologic drug therapy (moisturising creams allowed) in the study area or light therapy within the preceding 2 weeks
* Use of oral steroids within 1 month prior to the study
* Use of concurrent medication e.g. medication that may interfere with the study related activities
* Factors suggesting low compliance with study procedures
* Possible allergy to ingredients in the study medications
* Pregnancy or breast feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-01; Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To study the compatibility of the skin with the new formulation in comparison to the reference medication. | 3 weeks
To study the effect of maintenance therapy with an emollient cream on the possible recurrence of atopic eczema. | Up to 6 months

SECONDARY OUTCOMES:
To study cosmetic acceptance of the corticosteroids | 3 weeks
To study the safety of corticosteroid treatment. | 3 weeks
To study the safety of maintenance treatment. | Up to 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Berit Berne, MD, Principal Investigator — Hudkliniken, Akademiska sjukhuset, Uppsala
Locations (5):
- Sweden (5):
  - Nacka hudmottagning, Nacka
  - Nacka närsjukhus, Nacka
  - Sophiahemmet, Stockholm
  - Hudkliniken, Danderyds sjukhus, Stockholm
  - Läkarhuset Vällingby, Vällingby